CLINICAL TRIAL: NCT07356063
Title: Effect of a Multicomponent Support Group on Self-Efficacy of Primary Caregivers of Children With Spinal Muscular Atrophy or Duchenne Muscular Dystrophy Enrolled in Treat-NMD Registry of Pakistan
Brief Title: Self-Efficacy Enhancement Using a Multicomponent Support Group for Caregivers of Children With DMD/SMA
Acronym: SEE-NMD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sara Khan, Doctor, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-11875-37040
Record Dates: First submitted 2026-01-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy (DMD); Spinal Muscular Atrophy (SMA)
Keywords: DMD; SMA; Self-Efficacy; Caregivers; Treat-NMD; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Atrophy, Spinal; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: Pre intervention: Baseline assessment of self efficacy scoring will be taken from each participant, where they will rate each item on a 5-point Likert scale, on Zoom call.
  Post intervention: After 2 months, the participants of each group will be contacted for post intervention scoring via Zoom call.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicomponent Support Group Intervention for Caregivers of Children with DMD or SMA (Experimental): Participants receive a structured, online multicomponent support group designed for primary caregivers of children with DMD or SMA enrolled in the Treat-NMD Registry of Pakistan. The intervention includes educational sessions, peer support discussions, and guidance from professionals in physiotherapy, respiratory care, occupational therapy, and psychosocial coping. Caregiver self-efficacy will be assessed before and after the intervention to measure changes associated with participation.
  Interventions: Behavioral: Multicomponent Support Group

INTERVENTIONS:
Behavioral: Multicomponent Support Group — A multifaceted strategy will be employed. Multiple groups will be created for SMA and DMD patients. Each group will include up to 10 patients caregivers, 1 neurologist, 1 pediatric neurologist, 1 physiotherapist, 1 nutritionist, 1 speech therapist, 1 occupational therapist, 1 epidemiologist and 1 Research Associate. Sessions with each group will integrate peer support, coaching to address the multifaceted needs of patients, and time for open questions and answer sessions with the group. The session with each group will be 1 hours duration. It will start with 5 minutes talk from each expert about the basic needs for SMA and DMD patients. Following the first session, after a few weeks gap, another similar 1 hour session will be conducted which will be open to care givers to ask questions off the specialists or other care givers. In between these 2 sessions, short videos or pictorial clips for care will be sent to the participants to re-enforce what they learnt from sessions.

SUMMARY:
The goal of this clinical trial is to learn if providing a multicomponent intervention improves the confidence of caregivers of children with DMD or SMA. The main question it aims to answer is:

Does this intervention increase their self-efficacy scores over 8 weeks time?

Researchers will compare scores at baseline (pre intervention) and after 8 weeks (post intervention)

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) and Duchenne Muscular Dystrophy (DMD) are severe neuromuscular disorders that significantly impact the lives of affected children and their families, placing immense pressure on primary caregivers who often experience diminished self-efficacy due to the complexities of caregiving. Both conditions necessitate specialized and time-consuming care, creating substantial challenges for caregivers.These challenges are compounded by the progressive nature of these diseases, which often leads to increased functional decline, discomfort, and respiratory dysfunction in affected children. The constant need for monitoring, administering medication, providing physical support, and managing medical equipment can be overwhelming and exhausting. The complex care requirements associated with SMA and DMD can also lead to social isolation, financial strain, and emotional distress for caregivers, effecting their overall quality of life and potentially reducing their confidence in their ability to manage their caregiving responsibilities. Therefore, understanding interventions that can bolster self-efficacy among primary caregivers of children with SMA or DMD is of paramount importance.

Self-efficacy, defined as an individual's belief in their capacity to execute behaviours necessary to produce specific performance attainments, plays a pivotal role in coping with chronic illnesses and their demanding care routines. When caregivers possess high self-efficacy, they are more likely to approach challenges with confidence, persevere through difficulties, and experience lower levels of stress and burnout. Conversely, low self-efficacy can result in feelings of helplessness, anxiety, and depression, which can ultimately compromise the quality of care provided to the child and their own well-being. Given the substantial impact of SMA and DMD on both the affected children and their caregivers, interventions aimed at enhancing self-efficacy are critical. One such intervention is participation in support groups, which provide caregivers with opportunities to share experiences, gain knowledge, and receive emotional support from others facing similar challenges. While traditional in-person support groups have been shown to be beneficial, they may not always be accessible to caregivers due to geographical limitations, time constraints, or transportation difficulties.

Online support groups have emerged as a promising alternative, offering convenience, accessibility, and anonymity, which may be particularly appealing to caregivers who are already burdened with numerous responsibilities and constraints. These online platforms can facilitate peer-to-peer support, professional guidance, and access to valuable resources, all from the comfort of one's own home. Furthermore, multicomponent support groups using online modalities can integrate various elements, such as educational videos, interactive discussions, and lectures by trained professionals like Neurologists, Nutritionists, Physiotherapists. These may be particularly effective in enhancing self-efficacy by addressing the multifaceted needs of caregivers. Considering the potential benefits of multicomponent support group for primary caregivers of children with SMA or DMD, and the increasing prevalence and duration of chronic illness, there is a need for array of supports for them.

This study is designed to evaluate the effect of a multicomponent support group on the self-efficacy of primary caregivers of children with SMA or DMD enrolled in the Treat-NMD registry of Pakistan. By examining the effect of this intervention, we hope to provide evidence-based recommendations for improving the well-being of caregivers and, ultimately, the quality of care for children with SMA and DMD. The findings from this study will have significant implications for healthcare providers, support organizations, and policymakers involved in the care of individuals with neuromuscular disorders and their families.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child diagnosed with SMA or DMD.
* Enrolled in the Treat-NMD registry- Pakistan.
* Access to a smart phone with internet connectivity.

Exclusion Criteria:

* Caregivers who are currently participating in another support group intervention.
* Caregivers who are unable to understand the language of communication (Urdu)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Efficacy Scores | Baseline and 8 weeks
  Change from Baseline in the Self-Efficacy Scores at 8 weeks. Care giver self efficacy tool is a 19-item self-report questionnaire adapted from the original validated scale developed for caregivers of individuals with DMD (DMD-CSES). The scale assesses caregiver self-efficacy across multiple domains of caregiving.
  Each item is rated on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree).
  Total scores range from 19 to 95, calculated by summing responses across all items.
  Higher scores indicate greater caregiver self-efficacy (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Nashit Irfan Aziz, MBBS, MSc, Principal Investigator — Aga Khan University; Sara Khan, MBBS, MD, Principal Investigator — Aga Khan University; Wardah Khalid, MBBS, MSc, PhD, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Treat-NMD is a global organisation that brings together a network of leading specialists, patient groups and industry representatives. This in turn aims to ensure preparedness for the trials and therapies of the future while also promoting best practice — https://www.treat-nmd.org/treat-nmd-registry-network/
- See also: The Muscular Dystrophy Registry of Pakistan has been setup with a goal to improve outcomes and quality of life in patients with muscular dystrophies and related neuromuscular disorders. The registry is currently recruiting patients with Duchenne/Becker M — https://mdrpakistan.com/